CLINICAL TRIAL: NCT05759676
Title: A Prospective, Multicenter Observational Study of Efficacy and Safety of Polymer-free Amphilimus-eluting Stent (Cre8™/Cre8™ EVO) in Patients With Coronary Artery Disease According to the Presence of Diabetes Mellitus
Brief Title: Efficacy and Safety of Polymer-free Amphilimus-eluting Stent According to the Diabetes
Status: Recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Diomedical (Unknown)
Responsible Party: Principal Investigator, Soon Jun Hong, Professor, Korea University Anam Hospital
Other Study IDs: CRE8DM
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cre8™/Cre8™ EVO drug-eluting stent — Patient with CAD who undergoing PCI with Cre8™/Cre8™ EVO drug-eluting stent

SUMMARY:
Drug-eluting stents (DES) have been found to reduce the rate of stent restenosis compared to bare metal stents (BMS), but the first generation DES caused an increase in stent thrombosis. The second generation DES, including the Cre8Evo stent, has been designed to address these issues. The Cre8Evo stent is made of cobalt chromium and releases the drug amphilimus into the vessel wall, which is quickly absorbed and then lost, creating a BMS-like form. The Cre8Evo stent does not contain polymers and does not induce an inflammatory response. It inhibits cdk2 and RhoA, reducing the proliferation and migration of vascular smooth muscle cells. In diabetic patients, the Cre8Evo stent showed superior results in suppressing late proliferation compared to conventional DES. The Cre8Evo stent has been found to be safe and effective in clinical studies, and it has a superior effect in the clinical course of diabetic patients compared to other stents. The purpose of the study is to evaluate the effectiveness and safety of the Cre8Evo stent in actual clinical practice, specifically comparing outcomes in patients with and without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or older

  * Patients who agreed to the research protocol and clinical follow-up plan, voluntarily decided to participate in this study, and gave written consent to the consent form ③ Patients who underwent coronary angioplasty by inserting Cre8™ or Cre8™ EVO stent for coronary artery disease for a lesion confirmed within the last 1 month

Exclusion Criteria:

* Patients with known hypersensitivity or contraindications to the following drugs or substances: heparin, aspirin, clopidogrel, amphilimus, cobalt chrome, stainless steel nickel, 316L metal, and contrast media If it can be controlled by pheniramine and pheniramine, registration is possible, but if there is known anaphylaxis, it is excluded.)

  * Pregnant women, lactating women, or women of childbearing age who are planning to become pregnant during the study period ③ Patients who are planning surgery to stop antiplatelet drugs within 12 months from registration

    * Patients whose remaining life expectancy is expected to be less than 1 year

      * Patients who visited the hospital due to cardiogenic shock and are predicted to have a low survival rate based on medical judgment ⑥ Subjects participating in medical device randomization research ⑦ Patients who underwent surgery using a stent other than Cre8™/Cre8™ EVO at the time of registration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with coronary artery disease who is undergoing percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure(Device-oriented composite endpoints) | 12 month
  composite of cardiac death, any myocardial infarction not clearly attributatble to a non-target vessel, and clinical indicated target lesion revascularization in patient with DM and non-DM

SECONDARY OUTCOMES:
patient-oriented composite endpoint | 12 month
  composite of all-cause mortality, any myocardial infarction, and any revascularization in patient with DM and non-DM
Incidence of all-cause mortality | 12 month
  Incidence of all-cause mortality in patient with DM and non-DM
Incidence of all-cause cardiac death | 12 month
  Incidence of all-cause cardiac death in patient with DM and non-DM
Incidence of all-cause non-cardiac death | 12 month
  Incidence of all-cause non-cardiac death in patient with DM and non-DM
Incidence of any myocardial infarction | 12 month
  Incidence of any myocardial infarction in patient with DM and non-DM
Incidence of any myocardial infarction not clearly attributatble to a non-target vessel | 12 month
  Incidence of any myocardial infarction not clearly attributatble to a non-target vessel in patient with DM and non-DM
Incidence of any revascularization | 12 month
  Incidence of any revascularization in patient with DM and non-DM
Incidence of target lesion revascularization | 12 month
  Incidence of target lesion revascularization in patient with DM and non-DM
Incidence of stent thrombosis | 12 month
  Incidence of stent thrombosis in patient with DM and non-DM
Lesion success rate | the day of procedure
  less than 50% of residual stenosis after all procedure in patient with DM and non-DM
Procedural success rate | 1 month
  composite of less than 50% of residual stenosis after all procedure, no in-hospital event including death, MI, revascularization in patient with DM and non-DM

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The subject identification information used in the study will be coded and managed so that personal identification is impossible. Documents and materials related to this study will be stored in a locked place designated by the research director. In accordance with Article 15 of the Enforcement Rules of the Bioethics and Safety Act, research-related records are planned to be kept for 3 years from the time the research is completed, and documents that have passed the retention period will be destroyed according to the relevant grounds.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code